CLINICAL TRIAL: NCT04254445
Title: The Effect of Personalized Custom Training Videos on Patient Engagement in Hospitalized Patients Undergoing Thoracocentesis
Brief Title: Use of Guidance Videos to Increase Engagement and Decrease Anxiety in Patients Undergoing Pleural Tap
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GistMed Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0009-19-TLV
Record Dates: First submitted 2020-01-05; First posted 2020-02-05 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pleural Effusion; Pleural Effusion, Malignant; Pleural Pleurisy Effusion
Keywords: Personalized video training; Thoracocentesis; Pleural tap
MeSH Terms: conditions — Pleural Effusion; Pleural Effusion, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training video arm (Experimental): Patients will watch a personalized custom training video, in addition to the standard explanation provided by the medical staff
  Interventions: Other: Personalized training video
- Verbal explanation arm (No Intervention): Patients will standard explanation about the procedure, provided by the medical staff

INTERVENTIONS:
Other: Personalized training video — Using a few demographic and medical details of the patients, provided by the medical staff, the video generator will create a 2-minute personalized custom video, suitable to the age, gender, language, and medical condition of the patients. No identifying information will be used, to protect patient's privacy.
  Arms: Training video arm

SUMMARY:
Patients planned to undergo a pleural tap will get verbal explanation or watch a personalized guidance video in addition to verbal explanation. Questionnaires will be filled to assess the effect of the video training on understanding, cooperation and anxiety.

DETAILED DESCRIPTION:
100 patients with pleural effusion, planned to undergo a diagnostic or therapeutic pleural tap, will be randomized to watch a personalized custom video training, explaining the procedure, in addition to the verbal explanation given by the medical staff, or to get the standard verbal explanation alone. Questionnaires regarding their understanding of the procedure, their feelings and the level of anxiety will be filled before and after the video/verbal explanation, and after the procedure. the study aims to check whether the video training provides better understanding of the procedure, increases cooperation and engagement and decreases anxiety.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in Internal medicine C and D, Tel-Aviv Sourasky Medical Centers
* Patients with pleural effusion, planned to undergo diagnostic or therapeutic pleural tap
* Patients who can read and understand the questions
* Patients who were interested in participating in the clinical trial and signed an informed consent form

Exclusion Criteria:

* Minors < 18 years of age
* Pregnant women
* Patients who cannot read and understand, at the discretion of the investigator
* Patients which their medical condition does not allow them to undergo the study procedure

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-16 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Fulfillment of need for information gap | 30 minutes
  Improvement of subjective self-assessment of the patient's need of information on the tap procedure following the explanation received, based on the short form of the Quality from Patient Perspective (QPP) measurement. The improvement in the intervention arm will be compared to the one of the control arm
Assessment of Anxiety | 30 minutes
  Delta of subjective self-assessment on his/her anxiety about the procedure, following the explanation received (using visual scale of 1-100, based on the Visual Analog Scale (VAS)). The reduction of anxiety in the intervention arm will be compared to the one of the control arm

SECONDARY OUTCOMES:
The need of an active role | 30 Minutes
  The patients will be asked to score whether the explanation allowed them the active role they needed, based on the Picker Patient Experience (PPE-15) Questionnaire. The score in the intervention arm will be compared to the one of the control arm
Confidence and Knowledge to take actions | 30 minutes
  The patient would be asked to score whether the information they received allowed them to understand what they should do next, based on the Patient Activation Measure (PAM) Questionnaire. The score in the intervention arm will be compared to the one of the control arm

CONTACTS AND LOCATIONS:
Overall Officials: Orit Neudorfer, MD, Study Director — GistMed Ltd.
Locations (1):
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No